CLINICAL TRIAL: NCT02567474
Title: Effect of Self Management Program Based on 5A Model on Clinical Status of Chronic Obstructive Pulmonary Disease
Brief Title: Effect of Self Management Program on Clinical Status of COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahvaz Jundishapur University of Medical Sciences (Other)
Responsible Party: Principal Investigator, maryam heidari, principal investigator, Ahvaz Jundishapur University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P-327
Record Dates: First submitted 2015-09-27; First posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: COPD
Keywords: chronic lung disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): no intervention
- intervention (Experimental): self management intervention based on 5A model
  Interventions: Behavioral: 5 A model

INTERVENTIONS:
Behavioral: 5 A model — self management program based on 5A model
  Other Names: self managment
  Arms: intervention

SUMMARY:
This study evaluates the effectiveness of self management programs based on 5A model on the lung function status, dyspnea and exercise tolerance in Chronic Obstructive Pulmonary Disease patients. Participants were randomly assigned to an intervention group or a control group. The control group were receiving standard practice care and the intervention group were receiving intervention in addition to standard practice care. The intervention content include implementation of a self management plan based on 5A model.

DETAILED DESCRIPTION:
5 A model implemented during a period of 12 weeks including 5 stags: assessment of behavior, beliefs and motivation of the patient (Assess); provide information about personal health risks and benefits of change (Advise); mutual contribution of patients and health care provider on setting realistic goals based on the patient's interest and confidence in their ability to change the behavior (Agree); help anticipate barriers and develop practical applications based on the identified patient's strategies, problem-solving techniques and social/environmental support (Assist) and specify plan for follow-up (Visits, Phone calls) and providing support in the course of follow up (Arrange).

ELIGIBILITY:
Inclusion Criteria:

* certified diagnosis of COPD with moderate or severe level by a pulmonologist according to GOLD criteria
* age range of 45-70 years
* BMI<30
* being literate
* having a strong understanding of the Persian language
* having a constant prescription drug regime
* not suffering from another serious and restrictive disease (such as major psychological disorder, neural disease, musca-skeletal disease, cancer, cardiac or angina attack in last month)

Exclusion Criteria:

* hospitalization during the intervention
* need to use of oxygen or spray during 6-minute walking test
* dealing with serious stress
* failure of patient to attend personal or group education session
* non-compliance with a practical program that was determined at monthly visits for intervention group

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
dyspnea severity measured by dyspnea Borg scale | 3 month
  dyspnea was measured by dyspnea Borg scale. This scale is visual tool ranging from 0(not dyspnea) to 10(maximum dyspnea).

SECONDARY OUTCOMES:
exercise tolerance rate | 3 month
  exercise tolerance was measured by Six Minutes Walking Test.in this test the distance that each patient was able to walk under standard condition in 6 minutes was measured by researchers.
lung function status measured by spirometry | 3 month
  lung function was measured by spirometry. Spirometry is a test that measures how an individual inhales or exhales volumes of air as a function of time
quality of life | 3 month
  quality of life was measured by SF-36 Questionnaire. It consisted of 36 questions that examine the eight quality of life dimensions, each question has a continuous quantitative scale from 0 to 100, in which higher scores indicate better situation.

CONTACTS AND LOCATIONS:
Overall Officials: maryam heidari, M.sc, Principal Investigator — Department of Nursing, School of Nursing and Midwifery, Ahvaz Jundishapur University of Medical Science, Ahvaz, Iran.